CLINICAL TRIAL: NCT00648167
Title: A Safety and Tolerability Study of Zerenex (Ferric Citrate) in Patients With End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Collaborators: Collaborative Study Group (CSG) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-201
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hyperphosphatemia; End-stage Renal Disease
Keywords: ESRD; end-stage renal disease; end stage renal disease; hemodialysis; dialysis; kidney failure; renal failure; kidney; renal; phosphate binder; phosphorus
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic; Renal Insufficiency | interventions — ferric citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KRX-0502 (ferric citrate) (Experimental): All patients will be switched from their current phosphate binder to Zerenex, and titrated to the maximum tolerated dose (up to about 12g/day) based on their serum phosphorus levels.
  Interventions: Drug: ferric citrate

INTERVENTIONS:
Drug: ferric citrate — ferric citrate will be provided as a 375mg capsule. Dosing and frequency are dependent on patient's serum phosphorus levels. Dosing will occur over the 28-day study.
  Other Names: KRX-0502

SUMMARY:
This study is to evaluates the safety and tolerability of Zerenex™ (ferric citrate) as a treatment for hyperphosphatemia in patients with End-Stage Renal Disease.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of Zerenex™ (ferric citrate) as a treatment for hyperphosphatemia in patients with End-Stage Renal Disease. These patients will be switched to Zerenex™ from their current high dose of phosphate binder and, based on their serum phosphorus levels, will be titrated up from 3.4g/day of Zerenex™ to maximum tolerated and safe doses of Zerenex™. Doses will be adjusted weekly, based on serum phosphorus levels, with the maximum dose administered being approximately 12g/day.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, nonlactating females
* Age > 18 years
* On thrice weekly hemodialysis for at least the previous 3 months prior to randomization
* Phosphorous levels ≥3.5mg/dL at Screening Visit
* On at least 12 tablets/capsules/day of calcium acetate (667mg), calcium carbonate (500mg), lanthanum carbonate (500mg), sevelamer hydrochloride (800mg or two 400mg tablets), or any combination of these agents
* Serum ferritin <1000micrograms/L and Transferrin Saturation (TSAT) <50%
* Willing to be discontinued from current phosphate binder(s) and initiated on Zerenex
* Willing and able to give informed consent

Exclusion Criteria:

* Parathyroidectomy within 6 months prior to Screening
* Actively symptomatic GI disease such as peptic ulcer disease, gastro esophageal reflux, diverticulosis, irritable bowel syndrome (treated asymptomatic is permitted)
* History of documented inflammatory bowel disease or erosive esophagitis
* Serum Phosphorus levels >10.0 mg/dL documented in the 3 monthly laboratories (done routinely in the dialysis unit) in the 3 months prior to the Screening Visit
* History of multiple drug allergies
* History of malignancy in the last 5 years (treated cervical or skin cancer may be permitted if approved by CCC)
* Previous intolerance to oral ferric citrate
* Absolute requirement for oral iron therapy
* Absolute requirement for Vitamin C (multivitamins [Neprocaps, Renaphro, etc.] allowed)
* Absolute requirement for calcium, magnesium, or aluminum containing drugs with meals
* Psychiatric disorder that interferes with the patient's ability to comply with the study protocol
* Inability to tolerate oral drug intake
* Planned surgery or hospitalization during the study (scheduled outpatient access surgery allowed)
* Any other medical condition that renders the patient unable to or unlikely to complete the study or that would interfere with optimal participation in the study or produce significant risk to the patient
* Receipt of any investigational drug within 30 days of randomization
* Inability to cooperate with study personnel or history of noncompliance

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-03; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia B Lewis, MD, Study Chair — Collaborative Study Group at the Nephrology Clinical Trials Center, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor — http://www.keryx.com

RESULTS

PARTICIPANT FLOW:
Groups:
- KRX-0502: Ferric Citrate
Period: Overall Study
Arm/Group | KRX-0502
Started | 55
Start Dose 4.5 g/Day | 34
Start Dose 6 g/Day | 21
Completed | 48
Not Completed | 7
Not completed — Adverse Event | 6
Not completed — unable to swallow tablets | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat
Groups:
- KRX-0502: Subjects in this group were initiated on a dose of 4.5 g/day (34 subjects) or 6.0 g/day (21 subjects) of KRX-0502 (ferric citrate)
Arm/Group | KRX-0502
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.46 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 50
  Puerto Rico | 5

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Serum Phosphorus Between Baseline (Day 0) and End of Treatment (Day 28)
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- KRX-0502 (Ferric Citrate): Patients starting dose of 4.5 grams per day (n=34) and those starting on 6.0 grams per day (n=21)- immediate roll over from previous phosphate binder(s)
Arm/Group | KRX-0502 (Ferric Citrate)
Number analyzed (Participants) | 55
mg/dL
  Baseline | 5.9 (1.4)
  Day 28 | 5.4 (1.4)

ADVERSE EVENTS:
Groups:
- KRX-0502: Subjects in this group were initiated on a dose of 4.5 g/day (34 subjects) or 6.0 g/day (21 subjects) of KRX-0502 (ferric citrate)
  Intent-to-Treat (ITT)
Arm/Group | KRX-0502
Serious Adverse Events (participants affected / at risk) | 4/55
Other Adverse Events (participants affected / at risk) | 46/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KRX-0502 (N=55)
Liver infection (Infections and infestations) | 1 (1)
Methicillin - susceptible staphylococcus aureus bacteremia (Infections and infestations) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Worsened congestive heart failure (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KRX-0502 (N=55)
Stool color abnormality (Gastrointestinal disorders) | 34
Diarrhea (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Bloating (Gastrointestinal disorders) | 4
Heartburn (Gastrointestinal disorders) | 4
Stomach pain or cramp (Gastrointestinal disorders) | 4
Increased appetite (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No